CLINICAL TRIAL: NCT02524821
Title: Randomized, Open-label, 4-Way Crossover Study Assessing the Effect of Gelesis100 on the Pharmacokinetics of Metformin, Administered Under Fasting and Fed Conditions
Brief Title: The Effect of Gelesis100 on the Pharmacokinetics of Metformin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gelesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GS-100-005
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Healthy Overweight Obese
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- drugs only, fasted (Active Comparator): 1 x 850 mg metformin tablet, under fasting conditions.
  Interventions: Drug: Metformin
- Gelesis100 plus drugs, fasted (Experimental): 3 x 0.75 g Gelesis100 capsules, followed 30 minutes later by the administration of 1 x 850 mg metformin tablet, under fasting conditions.
  Interventions: Device: Gelesis100; Drug: Metformin
- drugs only, fed (Active Comparator): 1 x 850 mg metformin tablet, followed by the ingestion of a high-fat, high-caloric meal.
  Interventions: Drug: Metformin
- Gelesis100 plus drugs, fed (Active Comparator): 3 x 0.75 g Gelesis100 capsules, followed by the ingestion of a high-fat, high-caloric meal, followed by the administration of 1 x 850 mg metformin tablet (fed conditions).
  Interventions: Device: Gelesis100; Drug: Metformin

INTERVENTIONS:
Device: Gelesis100 — 3 capsules each containing 0.75 mg
  Arms: Gelesis100 plus drugs, fasted; Gelesis100 plus drugs, fed
Drug: Metformin — 1 tablet of 850 mg
  Other Names: Glucophage

SUMMARY:
The purpose of this study is to determine the effect of Gelesis100 on the absorption of metformin both with and without a meal.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco products within 3 months prior to screening), ≥ 22 and ≤ 65 years of age, with BMI ≥ 25.0 and ≤ 40.0 kg/m2.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to the first dosing (dosing refers to the administration of Gelesis100 or the substrate drugs, whichever comes first). Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Qualified Investigator.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
   3. the absence of history of lactic or metabolic acidosis.
   4. the absence of clinically significant history of gastric or peptic ulcer.
   5. the absence of clinically significant history or known presence of esophageal anatomic abnormalities (e.g., webs, diverticuli, rings), malabsorption, and gastroparesis.
   6. the absence of history of gastric bypass, any other gastric surgery and intragastric balloon.
3. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive method throughout the study and for 30 days after the last medical device/substrate drug administration:

   1. intra-uterine contraceptive device without hormone release system placed at least 4 weeks prior to medical device/substrate drug administration;
   2. condom with intravaginally applied spermicide starting at least 14 days prior to medical device/substrate drug administration.
4. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen or urine cotinine test at screening.
3. History of allergic reactions to metformin, carboxymethylcellulose, citric acid, sodium stearyl fumarate, raw cane sugar, gelatin, titanium dioxide, or other related drugs or substances.
4. Positive pregnancy test at screening.
5. Breast-feeding.
6. Any reason which, in the opinion of the Qualified Investigator, would prevent the subject from participating in the study.
7. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
8. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
9. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within 1 year prior to screening.
10. Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days (90 days for biologics) prior to the first dosing or concomitant participation in an investigational study involving no drug administration.
11. Use of medication other than topical products without significant systemic absorption:

    1. prescription medication within 14 days prior to the first dosing;
    2. over-the-counter products including natural health products (e.g., food supplements and herbal supplements) within 7 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
    3. a depot injection or an implant of any drug within 3 months prior to the first dosing.
12. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL within 30 days, or more than 499 mL within 56 days prior to the first dosing.
13. Hemoglobin <128 g/L (males) and <115 g/L (females) and hematocrit <0.37 L/L (males) and <0.32 L/L (females) at screening.
14. Subject with a small appetite or who would have difficulty to complete a high-fat, high-caloric meal, or to drink a large amount of liquid.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Effect of Gelesis100 on area under the curve (AUC) for plasma concentration of metformin under fed and fasted conditions | 0.5 to 24 hours post single dose (19 blood samples)
Effect of Gelesis100 on maximum plasma concentration (Cmax) of metformin under fed and fasted conditions | 0.5 to 24 hours post single dose (19 blood samples)
Effect of Gelesis100 on time to maximum plasma concentration (Tmax) of metformin under fed and fasted conditions | 0.5 to 24 hours post single dose (19 blood samples)

CONTACTS AND LOCATIONS:
Overall Officials: Audet, Principal Investigator — Quebec City, Quebec Canada
Locations (1):
- Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No